CLINICAL TRIAL: NCT05150444
Title: Effects of Intradialytic Cognitive and Physical Exercise Training on Functional Status of Hemodialysis Patients: Randomized Interventional Trial
Brief Title: Effects of Intradialytic Cognitive and Physical Exercise Training on Functional Status of Hemodialysis Patients
Acronym: DIAKOG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Špela Bogataj, Postdoctoral Researcher, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Z3-3212
Record Dates: First submitted 2021-11-25; First posted 2021-12-09 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Cognitive Dysfunction; Physical Inactivity; Chronic Kidney Diseases
Keywords: cognitive functions; hemodialysis; physical activity; intradialytic training; non-pharmacological interventions
MeSH Terms: conditions — Cognitive Dysfunction; Sedentary Behavior; Renal Insufficiency, Chronic; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive and physical exercise training (Experimental): This group will perform combined intradialytic cognitive and physical exercise training. First, they will exercise during dialysis (3 times a week; 12 weeks) for ~30 minutes on a customized ergometer. They will start with a 3-min warm-up, then the resistance will be implied to each individual according to the rate of perceived exertion of 4th to 5th grade on a 10-grade Borg scale. After a break, they will be given tablet computers in order to play "brain games" on a CogniFit platform (~30 - 45 min).
  Interventions: Other: Cognitive and physical exercise training
- Standard care (No Intervention): This group will receive standard hemodialysis care.

INTERVENTIONS:
Other: Cognitive and physical exercise training — 12 weeks (3 times a week): patients will cycle on an adapted ergometer during their dialysis procedure. The exercise program will be run by kinesiologists. Participants will start with 15 minutes of cycling and then gradually increase the time and intensity. After the physical exercise session, they will continue with cognitive training. This training will be done on a tablet computer on a CogniFit platform (~30 minutes). The "brain games" on mentioned platform automatically adapt to individual cognitive abilities.
  Arms: Cognitive and physical exercise training

SUMMARY:
The aim of this study is to investigate the effect of cognitive training combined with physical exercise on cognitive function, physical performance and frailty indicators in the hemodialysis population.

DETAILED DESCRIPTION:
The prevalence of cognitive impairment in hemodialysis (HD) patients is extremely high. Despite the well-documented benefits of interventions on cognitive function, there is a widespread call for effective strategies that will show the long-term consequences in patients undergoing dialysis. A randomized controlled intervention trial to examine the effects of a combined non-pharmacological intervention in the form of intradialytic physical exercise and intradialytic cognitive training on cognitive function, indicators of frailty, and physical performance measures in HD patients will be conducted. The group of patients receiving the study intervention will be compared to the control group receiving standard HD care. The duration of the intervention will be 12 weeks (3 days a week). We will use sensitive instruments (cognitive domain tests) to assess cognitive functions. The primary outcome of the study at 12 weeks will be performance on the Alertness subtest of the computerized Test of Attentional Performance. Secondary study outcomes will be: Performance in other domains of cognitive function (executive function, psychomotor speed, information processing efficiency, working memory, attention), physical fitness (10 repetition sit-to-stand test, timed up and go test, handgrip strength test, spontaneous gait speed, Stork balance test), and assessment of frailty (Edmonton Frail Scale). Study outcomes will be assessed at baseline and immediately after the 12-week intervention. This study will be among the first to test the synergistic effects of a uniquely designed physical exercise and cognitive training intervention on functional status in HD patients.

ELIGIBILITY:
Inclusion Criteria:

* dialysis patients on renal replacement therapy with chronic hemodialysis
* duration of hemodialysis treatment for at least 3 months
* capable of independent walking and independent feeding

Exclusion Criteria:

* the presence of chronic malignant or infectious disease
* uncontrolled arterial hypertension with an average of the last five pre-dialysis blood pressure values above 180/100 mm Hg,
* unstable angina pectoris or Canadian Cardiovascular Society class 2-4,
* heart failure New York Heart Association class 3 and 4,
* the presence of a psychotic illness or a mental disability,
* a condition with an amputated limb (more than 2 fingers on the lower limb and / or more than 2 fingers on the upper limb)
* any other condition that causes the clinical unstability of the patient (i.e. repetitive gastrointestinal hemorrhagies, liver cirrhosis with frequent exacerbations)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2022-11-02 (Actual); Primary Completion 2023-01-25 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Test of Attentional Performance (TAP) score | baseline, after 12 weeks
  The Test of Attentional Performance (TAP) is a software package that can be used primarily to examine attention functions. The rationale for the selection of the main outcome: low learning effect, most probably affected by physical exercise, attention is one of the most affected cognitive domains in dialysis patients. From the TAP test battery, subtests Alertness, Selective attention, and Divided attention will be included.

SECONDARY OUTCOMES:
Change in Montreal Cognitive Assessment (MoCA) score | baseline, after 12 weeks
  Montreal Cognitive Assessment (MoCA) is a global cognitive function assessment tool covering eight cognitive domains and is used to screen patients for cognitive impairment.
Change in Trail Making Test A and B score | baseline, after 12 weeks
  The psychomotor speed and executive function will be measured by Trail Making Test A and B.
Change in Symbol Digit Modalities Test (SDMT) score | baseline, after 12 weeks
  Symbol Digit Modalities Test (SDMT) will be used to assess the psychomotor speed, efficiency of information processing, ability to switch between mental sets of the information and to maintain and manipulate information in working memory. It is a reliable and valid test for assessing information processing speed and efficiency and executive functioning domains.
Change in 10 repetition sit-to-stand test time | baseline, after 12 weeks
  Performance of the sit-to-stand test involves activation of the lower limb muscles; the test measures lower limb strength. Participants are required to 10 times stand up from and sit down on an armless chair as quickly as possible. Their arms should be folded across their chest.
Change in Stork balance test time | baseline, after 12 weeks
  Stork balance test time as a measure of balance.
Change in frailty score | baseline, after 12 weeks
  Frailty indicator will be assessed by the Edmonton Frail Scale (EFS). The EFS score ranges from zero to 17 points. Severe Frailty is defined as a score of 12-17 possible points; apparent vulnerability is a score of 6-11 points; and non-frail is a score of 5 or less points.
Change in timed-up-and go (TUG) test time | baseline, after 12 weeks
  The Timed Up and Go (TUG) test is a simple evaluative test used to measure functional mobility. It will be used to estimate risk of falling and ability to maintain balance while walking and while walking and talking (TUG-dual).
Change in handgrip strength (HGS) test | baseline, after 12 weeks
  Handgrip strength test as a measure of upper body strength (in kilograms).
Change in Kidney Disease Quality of Life Short Form (KDQoL-SF) score | baseline, after 12 weeks
  Kidney Disease Quality of Life Short Form (KDQOL-SF) as a measure of quality of life. The scoring procedure first transforms the raw precoded numeric values of items to a 0-100 possible range, with higher transformed scores always reflecting better quality of life. Scores are evaluated according to summary scores: a mental component summary (MCS) and a physical component summary (PCS).
Change in spontaneous gait speed | baseline, after 12 weeks
  Spontaneous gait speed test (4 meters) as a measure of functional mobility (in m/s).
Change in Brain-derived neurotrophic factor (BDNF) concentration | baseline, after 12 weeks
  BDNF is a neurotrophic protein that promotes neurons' survival and differentiation.
Change in Interleukin-6 concentration | baseline, after 12 weeks
  Interleukin-6 serum concentration
Change in C-reactive protein (CRP) concentration | baseline, after 12 weeks
  C-reactive protein serum concentration
Change in hemoglobin concentration | baseline, after 12 weeks
  Hemoglobin blood concentration
Change in urea concentration | baseline, after 12 weeks
  Urea serum concentration
Change in phosphate concentration | baseline, after 12 weeks
  Phosphate serum concentration
Change in albumin concentration | baseline, after 12 weeks
  Albumin serum concentration
Change in fat tissue index | baseline, after 12 weeks
  Fat tissue index measured by bioimpedance analysis (BCM Fresenius Medical Care)
Change in lean tissue index | baseline, after 12 weeks
  Lean tissue index measured by bioimpedance analysis (BCM Fresenius Medical Care)
Change in mental fatigue | baseline, after 12 weeks
  Mental fatigue measured by Visual Analogue Scale (M-VAS) ranged 0-100, where higher score indicates higher mental fatigue.
Change in hematocrit concentration | baseline, after 12 weeks
  Hematocrit blood concentration
Change in creatinine concentration | baseline, after 12 weeks
  Creatinine serum concentration
Change in sodium concentration | baseline, after 12 weeks
  Sodium serum concentration
Change in potassium concentration | baseline, after 12 weeks
  Potassium serum concentration

CONTACTS AND LOCATIONS:
Overall Officials: Jadranka Buturović Ponikvar, PhD, Study Chair — University Medical Centre Ljubljana
Locations (1):
- University Medical Centre, Ljubljana, Osrednjeslovenska, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bogataj S, Trajkovic N, Pajek M, Pajek J. Effects of Intradialytic Cognitive and Physical Exercise Training on Cognitive and Physical Abilities in Hemodialysis Patients: Study Protocol for a Randomized Controlled Trial. Front Psychol. 2022 Jan 25;13:835486. doi: 10.3389/fpsyg.2022.835486. eCollection 2022. PMID 35145465